CLINICAL TRIAL: NCT01419470
Title: Phase Ⅰ/Ⅱ Clinical Trial to Investigate the Safety, Tolerability, Pharmacokinetics and Efficacy of YHD1044 After Oral Administration in Premature Ejaculation Patients
Brief Title: Safety, Tolerability, Pharmacokinetics and Efficacy of YHD1044
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Yuhan Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: YCD173
Record Dates: First submitted 2011-06-09; First posted 2011-08-18 (Estimated); Last update posted 2012-08-01 (Estimated); Status verified 2012-07

CONDITIONS: Premature Ejaculation
MeSH Terms: conditions — Premature Ejaculation | interventions — dapoxetine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- YHD1044 I (Experimental)
  Interventions: Drug: dapoxetine
- YHD1044 III (Experimental)
  Interventions: Drug: dapoxetine
- YHD1044 V (Experimental)
  Interventions: Drug: dapoxetine

INTERVENTIONS:
Drug: dapoxetine — 1. multiple dosing
  2. 12 subjects will be administered YHD1044 (I, III, V) or active/placebo comparators;dapoxetine
  Other Names: Priligy

SUMMARY:
safety and tolerability, pharmacokinetics/efficacy of an escalating, repeat doses of YHD1044 in premature ejaculation

ELIGIBILITY:
Inclusion Criteria:

* Patient is in a stable, monogamous sexual relationship with the same woman for at least 6 months and plans to maintain this relationship for the duration of the study
* History of premature ejaculation in the 6 months before study initiation
* History of intravaginal ejaculatory latency time (IELT) of < = 2 minutes in at least half of events
* Premature Ejaculation Diagnostic Tool (PEDT) > =11
* 6 domains of International Index of Erectile Function(IIEF) >= 21
* Patient and partner must agree to attempt sexual intercourse at minimum intervals specified in the protocol
* Patient's partner must have a negative urine pregnancy test at time of screening

Exclusion Criteria:

* Medical history which affects ADME in the past 3 years
* Clinically significant and active disorder in ophthalmic system, gastro-intestine, cardiovascular, respiratory system, endocrine system, autoimmune system or malignant tumor,
* Subjects with clinically significant observations considered as unsuitable based on medical judgment in the physical examination and clinical laboratory tests or a medical history
* History of psychological disease
* Clinically significant allergic disease
* Hypersensitivity to TCA, SSRIs(Clomipramine, sertraline, fluoxetine, dapoxetine)
* Taken dapoxetine within 3 months
* Using other forms of therapy for treatment of PE (behavioral therapy or medications applied to the skin)
* Taken another investigational drug within 1 month
* History of drug abuse

Ages: 20 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2011-02; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability | throughout the study up to day 28
  through physical examination, laboratory result, vital sign,ECG etc.

SECONDARY OUTCOMES:
Efficacy(IELT) | 13days, 28days
  change from baseline in IELT at the Day 13, 28
Cmax(Cmax,ss), Cmin,ss, AUCinf, AUCt, Tmax, CL/F | specified timepoints in the protocol
  Cmax(Cmax,ss), Cmin,ss, AUCinf, AUCt will be assessed. Samping time point: intensive sampling(Day1~2, Day14~15)& intermittent sampling(Day3~Day 28 except intensive sampling period)

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung medical center, Seoul, Seoul, South Korea